CLINICAL TRIAL: NCT03330067
Title: Warm and Humidified vs Cold and Dry Dry Carbon Dioxide (CO2) Pneumoperitoneum in Minimally Invasive Colorectal Resection: A Randomized Controlled Trial and Study of Clinical Endpoints
Brief Title: Warm and Humidified vs Cold and Dry Carbon Dioxide (CO2) Pneumoperitoneum
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are not performing the study and we don't plan to continue. We do not have support to complete the study.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 16-2223
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pneumoperitoneum
Keywords: laparoscope
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Before surgery patients will be assigned to one of two types of CO2 gas (conventional-room temperature and dry, or conditioned-95°F and 95% humidity) by a method similar to the flip of a coin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cold and dry CO2 pneumoperitoneum (Sham Comparator): Pneumoperitoneum is created by insufflation of standard cold (19-21°C) and nonhumidified (0%) CO2 directly from a standard CO2 tank or wall source.
  Interventions: Device: Cold and dry CO2 pneumoperitoneum
- Warm and humidified CO2 pneumoperitoneum (Experimental): The humidification and warming device to be used is the Insuflow Synergy Port (Lexion Company, FDA approved) which is a specialized 5 mm port that delivers warmed (95° F) and humidified (95% relative humidity) CO2, the source of which is a standard CO2 tank or wall source.
  Interventions: Device: Warm and humidified CO2 pneumoperitoneum

INTERVENTIONS:
Device: Cold and dry CO2 pneumoperitoneum — In this arm, patients undergo pneumoperitoneum by the insufflation of cold (19-21°C) and nonhumidified (0%) CO2.
  Arms: Cold and dry CO2 pneumoperitoneum
Device: Warm and humidified CO2 pneumoperitoneum — In this arm, patients undergo pneumoperitoneum by the insufflation of warmed (95° F) and humidified (95% relative humidity) CO2, using a Lexion Insuflow device.
  Other Names: Lexion Insuflow device
  Arms: Warm and humidified CO2 pneumoperitoneum

SUMMARY:
Laparoscopic surgery (surgery with the use of a camera and small instruments) uses insufflation, which is the standard medical practice where CO2 (carbon dioxide) gas is blown into the abdomen to create space for surgical procedures. The purpose of this study is to investigate whether heating and humidifying surgical CO2 will reduce surgery-related inflammation and postoperative pain.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial in which 120 patients undergoing elective laparoscopic colorectal resection will either undergo insufflation of the peritoneum with cold and dry (CD), control or warm and humidified (WH) CO2, experimental. Patients scheduled to undergo elective Laparoscopic Colon Resection (LCR) will be informed about the study and all questions answered. Consenting patients will be randomized (via envelope system) to have either standard cold (19-21°C) and nonhumidified (0%) CO2 or warm (37°C) and humidified (95%) CO2 utilized for their resection. To ensure that similar numbers of rectal resection patients are in each group, a separate envelop randomization will be used for colectomy and rectal resection cases.

The study will be conducted at Mount Sinai West hospital. The ambient operating room temperature will be regulated to 70-72° F. All patients will undergo laparoscopic surgery. During laparoscopic surgery the camera and instruments are inserted into the abdomen via small incisions allowing for the surgeon to explore the whole abdominal cavity without making larger cuts. In order to create space for surgical procedures, insufflation with CO2 is used. Regarding the method of insufflation, subjects will be randomized into 2 groups: i) standard CD CO2 insufflation ii) Lexion Insuflow device providing warmed humidified CO2 insufflation (95° F and 95% relative humidity) The humidification and warming device to be used is the Insuflow Synergy Port (Lexion Company, FDA approved) which is a specialized 5 mm port that delivers warmed (95° F) and humidified (95% relative humidity) CO2, the source of which is a standard CO2 tank or wall source. This study was conceived and designed by the PI who approached Lexion seeking devices for the study. The company will provide no funds for the study and the data and all decision regarding presentation and publications are to be made by Mount Sinai West research team.

Study patients will receive anesthesia according to the following regimen (Mount Sinai West anesthesia department has suggested this regimen and has agreed to abide by it for LCR patients unless there is a contraindication to this approach in a given patient): Induction anesthesia will include IV midazolam, IV fentanyl (3-5 mcg/kg), IV propofol, IV rocuronium, perioperative IV antibiotics, IV ondansetron for nausea prophylaxis, IV dexamethasone (8mg), IV acetaminophen 1000mg, and IV ketorolac 15 mg. Maintenance anesthesia will included IV fentanyl (1-2 mcg/kg/hr), sevoflurane or desflurane inhalational agent, and 100% oxygen. Fentanyl doses can be increased at the discretion of the anesthesiologist. 30-40 minutes before the end of the procedure, the intraoperative narcotics will be discontinued and hydromorphone PCA will be started. Patients will receive hydromorphone in the post anesthesia care unit according to the discretion of the anesthesiologist.

Analysis: Data will be recorded by the Study RN and/or the research resident on a daily basis on Case Report Forms (paper) which will be entered into a HIPPA compliant dedicated study data base with access limited to study personnel and our data manager. The Non-parametric and parametric tests such as Kruskal-Wallis test and Analysis of Variance test shall be used to determine the impact of warm humidified vs cold dry CO2 on postoperative pain medication requirements as well as on other operative and short term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic colorectal resection (LCR) for all indications (cancer, diverticular disease, benign neoplasm, inflammatory bowel disease, etc)

Exclusion Criteria:

* Patients younger than 18 and older than 85, emergency surgery, reoperation within 30 days, patients who are taking pain medications (either NSAID's or narcotics) on a daily basis preoperatively for whatever reason, patients with a history of narcotics addiction, paraplegic and quadriplegic patients, patients with dementia or altered mental status, and patients on steroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of pain medications taken postoperatively | up to 7 days
  The number of pain medications administered while hospitalized postoperatively will be tracked and recorded.
Timing of pain medications taken postoperatively | up to 7 days
  The timing of pain medications administered while hospitalized postoperatively will be tracked and recorded.

SECONDARY OUTCOMES:
Postoperative pain levels | up to 21 days
  Postoperatively, pain levels (visual analog hospital pain scale) will be measured and recorded. scale from no pain (0) to worse pain (10).
Number of pain medications taken after discharge | up to 21 days
  Patients will likewise record the type and number of pain medications taken after discharge.
Intraoperative narcotic use | Day 1
Analgesia requirements in the post anesthesia care unit | Day 1
Volume of CO2 consumed during surgery | Day 1
  CO2 gas volumes required for LCR
Length of stay | up to 21 days
Time to first flatus | up to 21 days
Time to first bowel movement | up to 21 days
Time to solid diet | up to 21 days
Postoperative complications | up to 21 days
Duration of Surgery | Day 1
Incision length | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whelan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuhaus SJ, Gupta A, Watson DI. Helium and other alternative insufflation gases for laparoscopy. Surg Endosc. 2001 Jun;15(6):553-60. doi: 10.1007/s004640080060. Epub 2001 Apr 3. PMID 11591939
- [Background] Brokelman WJ, Lensvelt M, Borel Rinkes IH, Klinkenbijl JH, Reijnen MM. Peritoneal changes due to laparoscopic surgery. Surg Endosc. 2011 Jan;25(1):1-9. doi: 10.1007/s00464-010-1139-2. Epub 2010 Jun 15. PMID 20552372
- [Background] Erikoglu M, Yol S, Avunduk MC, Erdemli E, Can A. Electron-microscopic alterations of the peritoneum after both cold and heated carbon dioxide pneumoperitoneum. J Surg Res. 2005 May 1;125(1):73-7. doi: 10.1016/j.jss.2004.11.029. PMID 15836853
- [Background] Holmdahl L, Ivarsson ML. The role of cytokines, coagulation, and fibrinolysis in peritoneal tissue repair. Eur J Surg. 1999 Nov;165(11):1012-9. doi: 10.1080/110241599750007810. PMID 10595602
- [Background] Almeida OD Jr. Awake microlaparoscopy with the Insuflow device. JSLS. 2002 Jul-Sep;6(3):199-201. PMID 12166755
- [Background] Demco L. Effect of heating and humidifying gas on patients undergoing awake laparoscopy. J Am Assoc Gynecol Laparosc. 2001 May;8(2):247-51. doi: 10.1016/s1074-3804(05)60585-3. PMID 11342732
- [Background] Jacobs M, Verdeja JC, Goldstein HS. Minimally invasive colon resection (laparoscopic colectomy). Surg Laparosc Endosc. 1991 Sep;1(3):144-50. PMID 1688289
- [Background] Braga M, Vignali A, Gianotti L, Zuliani W, Radaelli G, Gruarin P, Dellabona P, Di Carlo V. Laparoscopic versus open colorectal surgery: a randomized trial on short-term outcome. Ann Surg. 2002 Dec;236(6):759-66; disscussion 767. doi: 10.1097/01.SLA.0000036269.60340.AE. PMID 12454514
- [Background] Chen HH, Wexner SD, Weiss EG, Nogueras JJ, Alabaz O, Iroatulam AJ, Nessim A, Joo JS. Laparoscopic colectomy for benign colorectal disease is associated with a significant reduction in disability as compared with laparotomy. Surg Endosc. 1998 Dec;12(12):1397-400. doi: 10.1007/s004649900867. PMID 9822465
- [Background] Franklin ME Jr, Rosenthal D, Abrego-Medina D, Dorman JP, Glass JL, Norem R, Diaz A. Prospective comparison of open vs. laparoscopic colon surgery for carcinoma. Five-year results. Dis Colon Rectum. 1996 Oct;39(10 Suppl):S35-46. doi: 10.1007/BF02053804. PMID 8831545
- [Background] Franklin ME Jr, Rosenthal D, Norem RF. Prospective evaluation of laparoscopic colon resection versus open colon resection for adenocarcinoma. A multicenter study. Surg Endosc. 1995 Jul;9(7):811-6. doi: 10.1007/BF00190088. PMID 7482191
- [Background] Schwenk W, Bohm B, Muller JM. Postoperative pain and fatigue after laparoscopic or conventional colorectal resections. A prospective randomized trial. Surg Endosc. 1998 Sep;12(9):1131-6. doi: 10.1007/s004649900799. PMID 9716766
- [Background] Birch DW, Manouchehri N, Shi X, Hadi G, Karmali S. Heated CO(2) with or without humidification for minimally invasive abdominal surgery. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD007821. doi: 10.1002/14651858.CD007821.pub2. PMID 21249696
- [Background] Ott DE, Reich H, Love B, McCorvey R, Toledo A, Liu CY, Syed R, Kumar K. Reduction of laparoscopic-induced hypothermia, postoperative pain and recovery room length of stay by pre-conditioning gas with the Insuflow device: a prospective randomized controlled multi-center study. JSLS. 1998 Oct-Dec;2(4):321-9. PMID 10036122